CLINICAL TRIAL: NCT02071316
Title: The Use of Hexacapron in Upper Gastrointestinal Bleeding
Acronym: HEXUGI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Dr Bernardo Melamud, Dr.Bernardo Melamud, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Hexacap - 1
Record Dates: First submitted 2014-02-18; First posted 2014-02-25 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Upper Gastrointestinal Bleeding; Hexacapron; Hemostasis; Rebleeding; Mortality
Keywords: upper gastrointestinal bleeding; Hexacapron; hemostasis
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group, hexacapron , esomeprazole (Active Comparator): Treatment group - receive I.V. esomeprazole 80 mg and 8mg/h continuously with concurrent hexacapron I.V. every 6 hours until 72 hours and then continue oral treatment 6 g /day for 7 days.
  Interventions: Drug: Hexacapron( Tranexamic acid)
- Standard of care group, esomeprazole (Placebo Comparator): * Standard of care group - receive I.V. esomeprazole 80 mg once then 8mg/h continuously
  Interventions: Drug: esomeprazole

INTERVENTIONS:
Drug: Hexacapron( Tranexamic acid) — 1. Treatment group - receive I.V. Esomeprazole 80 mg once and then 8mg/h continuously with concurrent hexacapron( Tranexamic acid) I.V. every 6 hours until 72 hours and then the patient continue oral treatment 6 g /day for 7 days.
  Arms: Treatment group, hexacapron , esomeprazole
Drug: esomeprazole — 2. Standard of care group - receive I.V. Esomeprazole 80 mg once and then 8mg/h continuously
  Arms: Standard of care group, esomeprazole

SUMMARY:
The purpose of this study is to conduct a randomized control trial, double-blind study to compare Hexacapron with standard of care treatment to standard of care alone to evaluate the efficacy of adding effect of Hexacapron to standard therapy by decreasing the episodes of rebleeding and mortality in patient with upper gastrointestinal bleeding.

DETAILED DESCRIPTION:
Research Objectives

To evaluate the efficacy of using hexacapron in treatment of upper gastrointestinal bleeding

* Primary outcome: Prevention of rebleeding manifested as hematemesis, melena and drop in hemoglobin level by 2g% within 24 hours after therapeutic endoscopy
* Secondary outcomes: rebleeding, need for surgery , 30 day mortality

Expected Significance- The sample size needed to detect a 10% absolute difference in the proportion of rebleeding, drop in hemoglobin by 2g% between the hexacapron treated group and standard of care group groups with 80% power and 0.05 significant levels(alpha).

Research methods:

* Prospective , randomized controlled trial , double blinded , single center
* Duration : 2 years
* ~ 300≤ participants ,18≤ years of age
* Patients 18≤ years of age admitted to emergency department in Shaare Zedek Medical Center with clinical signs and symptoms of upper gastrointestinal bleeding will receive initial resuscitation and stabilization maintaining blood pressure and intravascular volume.

Patients will be randomized to 3 groups:

1. Treatment group - receive I.V. Esomeprazole 80 mg once and then 8mg/h continuously with concurrent hexacapron I.V. every 6 hours until 72 hours and then the patient continue oral treatment 6 g /day for 7 days.
2. Standard of care group - receive I.V. Esomeprazole 80 mg once and then 8mg/h continuously

   * Every patient will undergo upper endoscopy within 12 hours of admission to emergency department and receive treatment according to the endoscopic findings
   * If no reason for bleeding will be found in upper endoscopy , treatment will be stopped and patient will be excluded
   * Every participant will fill a questionnaire with informed consent which will have to be signed.

     * If cannot sign due to his medical condition or disability his guardian will sign or first degree relative

Study population:

Patients 18≤ years of age admitted to emergency department in Shaare Zedek MedicalCenter with clinical signs and symptoms of upper gastrointestinal bleeding including hematemesis, melena and drop in hemoglobin level by 2g%

Included:

* Patients 18≤ years of age admitted to emergency department in Shaare Zedek Medical Center with clinical signs, symptoms and laboratory of upper gastrointestinal bleeding
* Hospitalized patients in Shaare Zedek Medical Center with clinical signs, symptoms and laboratory of upper gastrointestinal bleeding • Patients , guardian or family member who can sign on informed consent

Excluded:

* Pregnancy, lactation
* History of thromboembolic event
* Allergic reaction to the drug
* Lower gastrointestinal bleeding
* Patient receive anticoagulation treatment
* Receive drug with interaction to hexacapron

ELIGIBILITY:
Inclusion Criteria:

* Patients 18≤ years of age admitted to emergency department in Shaare Zedek MedicalCenter with clinical signs, symptoms and laboratory of upper gastrointestinal bleeding
* Hospitalized patients in Shaare Zedek Medical Center with clinical signs, symptoms and laboratory of upper gastrointestinal bleeding
* Patients , guardian or family member who can sign on informed consent

Exclusion Criteria:

Pregnancy, lactation

* History of thromboembolic event
* Allergic reaction to the drug
* Lower gastrointestinal bleeding
* Patient receive anticoagulation treatment
* Receive drug with interaction to hexacapron

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Prevention of rebleeding manifested as hematemesis, melena and drop in hemoglobin level by 2g% within 24 hours after therapeutic endoscopy | Will be assessed 48 hours after admission to hospital
  All patients will undergo upper endoscopy within 12 hours from admission to assess their cause of upper GI bleeding .Patients will be evaluated according to the intervention group or standard of care group if there is another episode of bleeding or not during the first 48 hours after the first bleeding episode or within 24 hours after the first endoscopy was done

SECONDARY OUTCOMES:
Rebleeding, need for surgery , 30 day mortality | will be assessed after 30 days from admission to hospital
  All patients will be assessed for more bleeding episodes (>2 episodes) , need fo surgery or mortality during the 30 days after the first bleeding episode

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel, Israel